CLINICAL TRIAL: NCT03220685
Title: Relationship Between Gut Microbiota And Anemia In Patients With Chronic Renal Faliure
Brief Title: Relationship Between Gut Microbiota And Anemia In Patients With Chronic Renal Failure
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Ismaiel, Principal Investigator, Assiut University
Other Study IDs: Amr abdelrady 123
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2021-10

CONDITIONS: Gut Micrbota and Its Relation to Anemia of CKD Patients
Keywords: Microbiota
MeSH Terms: interventions — Occult Blood

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1.normal persons: normal persons include 25 person
  Interventions: Biological: Stool analysis
- 2.CKD pt with anemia: includes 25 previously diagnosed CKD patients with or without treatment of anemia.

INTERVENTIONS:
Biological: Stool analysis — Bacterial extraction in faeces by repeated fractional centrifugation to obtain bacterial mass and DNA sequencing.
  Groups: 1.normal persons

SUMMARY:
The human intestinal tract harbours a diverse and complex microbial community which plays a central role in human health. It has been estimated that our gut contains in the range of 1000 bacterial species and 100-fold more genes than are found in the human genome . This community is commonly referred to as our hidden metabolic 'organ' due to their immense impact on human wellbeing, including host metabolism, physiology, nutrition and immune function. It is now apparent that our gut microbiome coevolves with us and that changes to this population can have major consequences, both beneficial and harmful, for human health. Indeed, it has been suggested that disruption of the gut microbiota (or dysbiosis) can be significant with respect to pathological intestinal conditions such as obesity and malnutritio, systematic diseases such as diabetes and chronic inflammatory diseases such as inflammatory bowel disease (IBD), encompassing ulcerative colitis (UC) and Crohn's disease (CD) .

The role of the gut microbiome in human health and disease is becoming clearer thanks to high throughput sequencing technologies (HTS) as well as parallel recent developments in non genomic techniques.

DETAILED DESCRIPTION:
From the early stages of chronic kidney disease (CKD) there is a quantitative and qualitative alteration of intestinal microflora (dysbiosis); so the composition and metabolic activities of microflora are changed in CKD. These alterations include changes in intestinal transit, decreased protein absorption, decrease in dietary fibre intake, treatment with oral iron and frequent use of antibiotics.

All of this contributes to systemic inflammation and the accumulation of uraemic toxins that are absorbed by intestine and eliminated by the kidney.

This uraemic toxins have been associated with deleterious biological effects in different tissues and cell lines and with an increased risk of the progression of CKD, morbidity and mortality)

* Progression of CKD: both indoxyl sulfate(IS) and p-cresyl sulfate (PCS) are associated to the development of fibrosis, deterioration of renal function and disease progression . In vitro studies have shown a deleterious effect of these molecules on renal tubular cells. - Cardiovascular complications: in CKD patients, IS is associated with endothelial damage, arterial stiffness and aortic calcification .
* Anaemia: IS has been associated with anaemia of the renal patient; it interfere with the adequate production of erythropoietin and increased eryptosis (programmed cell death of red blood cells) .Polyamines are associated to anaemia in renal patients, through an intra-erythrocytic effect ,reduces erythropoiesis, and inhibit the activity of erythropoietin)
* Alterations of bone-mineral metabolism: IS reduces bone formation by promoting oxidative stress in osteoblasts and inducing resistance to PTH, which favours the development a dynamic bone .There is a positive correlation between FGF-23 and IS serum levels, suggesting an association between this molecule and metabolic bone disease in uraemic patients .
* Insulin resistance: In CKD patients the catabolism of insulin is reduced and often, they also have insulin resistance, which is associated with an increased risk of mortality; it seems that insulin resistance is related to some of the uremic toxins .

ELIGIBILITY:
Inclusion Criteria:

1 - Subjects participating in this study are CKD patients having eGFR less than 60 mL/min/1.73m2 for more than three months.

2. Individuals may be taking laxative drugs but they must be discontinued 3or more weeks before admission.

3. Age 18-70 years (in order to minimize the effect of aging on gut microbiota).

Exclusion Criteria:

* Subjects with a history or clinical manifestation of:

  1. Gastrointestinal disease, including inflammatory bowel diseases (e.g. Crohn s disease and ulcerative colitis), malabsorption syndromes (e.g. celiac disease), gastric ulcer (active) and irritable bowel syndrome.
  2. Lactose intolerance.
  3. Eating disorders such as anorexia nervosa , bulimia and binge eating syndrome.
  4. Taking weight loss drugs.
  5. Use of any antibiotic or probiotic agents within 6 months prior to minimize the potential effects of these substances on the gut microbiota.
  6. Use of antacids (Proton pump inhibitors, H2 antagonists or aluminum/magnesium hydroxide) 3 months prior to the study assessed by self-report because a modified gastric pH might affect the gut microbiota as well.
  7. Evidence of alcohol and/or drug abuse (more than 3 drinks per day and use of drugs, such as amphetamines, cocaine, heroin, or marijuana).
  8. Diabetic patients.
  9. Patients on dialysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To all patients history and clinical examination will be done plus routine investigation will be also done.
  Laboratory and imaging evaluation, as following:-
  1. Complete blood count
  2. serum creatinin and eGFR.
  3. Bacterial extraction in faeces by repeated fractional centrifugation to obtain bacterial mass and DNA sequencing.
  4. H.Pylori Ag in stool.
  5. Iron studies (TSAT).
  6. Abdominal ultrasound.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Relationship Between Gut Microbiota And Anemia In Chronic Kidney Disease (CKD) patients | 2 years
  1. Identifying dysbiosis and its role in anemia of CKD patients.
  2. Targeting of specific components of the gut microbiome of CKD patients and their correlation with anemia.
  3. To identify the effect of treatment of anemia with erythropoietin and iron therapy in CKD patients on the gut microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Kamal, Dr, Principal Investigator — Lecturer
Locations (1):
- Assiut universitu, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No